CLINICAL TRIAL: NCT01097746
Title: A Phase II Trial of Bevacizumab With Carboplatin and Weekly Paclitaxel as First-Line Treatment in Epithelial Ovarian, Primary Peritoneal, and Fallopian Tube Carcinoma
Brief Title: First-Line Treatment of Bevacizumab, Carboplatin, and Paclitaxel in Treating Participants With Stage III-IV Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0186; NCI-2018-01832 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0186 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Results first posted 2022-06-10 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-09

CONDITIONS: Fallopian Tube Carcinoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; FIGO Stage III Ovarian Cancer; FIGO Stage IIIA Ovarian Cancer; FIGO Stage IIIA1 Ovarian Cancer; FIGO Stage IIIA1(i) Ovarian Cancer; FIGO Stage IIIA1(ii) Ovarian Cancer; FIGO Stage IIIA2 Ovarian Cancer; FIGO Stage IIIB Ovarian Cancer; FIGO Stage IIIC Ovarian Cancer; FIGO Stage IVA Ovarian Cancer; FIGO Stage IVB Ovarian Cancer; Malignant Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Carcinoma; Primary Peritoneal Serous Adenocarcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Brenner Tumor | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (paclitaxel, carboplatin, bevacizumab) (Experimental): Participants receive paclitaxel IV over 3 hours on days 1, 8 and 15 and carboplatin IV over 1 hour on day 1. Beginning course 2, participants also receive bevacizumab IV over 1.5 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II trial studies how well first-line treatment of bevacizumab, carboplatin, and paclitaxel work in treating participants with stage III- IV ovarian, primary peritoneal and fallopian tube cancer. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving bevacizumab, carboplatin, and paclitaxel as first-line treatment may work better at treating ovarian, primary peritoneal, and fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether patients with newly diagnosed ovarian, primary peritoneal, and fallopian tube cancers when treated with bevacizumab, carboplatin, and weekly paclitaxel can tolerate at least 4 cycles of therapy regardless of delay or dose modification.

SECONDARY OBJECTIVES:

I. To estimate the efficacy of bevacizumab combined with carboplatin and weekly paclitaxel in patients with newly diagnosed ovarian, primary peritoneal, and fallopian tube cancers, as measured by progression-free survival.

II. To evaluate the response rate in patients with newly diagnosed ovarian, primary peritoneal, and fallopian tube cancers when treated with bevacizumab, carboplatin, and weekly paclitaxel.

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To assess the predictive value of a set of angiogenic genes whose expression correlates with progression-free survival of patients with epithelial ovarian, peritoneal primary or fallopian tube cancer treated with bevacizumab, carboplatin, and weekly paclitaxel.

II. To assess the relationship among cytokines/chemokines, angiogenesis factors, novel targets of interest and clinical outcome including tumor response and progression-free survival in patients treated with bevacizumab, carboplatin, and weekly paclitaxel.

OUTLINE:

Participants receive paclitaxel intravenously (IV) over 3 hours on days 1, 8 and 15 and carboplatin IV over 1 hour on day 1. Beginning course 2, participants also receive bevacizumab IV over 1.5 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologic diagnosis of epithelial ovarian cancer, peritoneal primary carcinoma or fallopian tube cancer; FIGO stage III and IV defined surgically at the completion of initial abdominal surgery and with appropriate tissue available for histologic evaluation. The minimum surgery required is an abdominal surgery providing tissue for histologic evaluation and establishing and documenting the primary site and stage, as well as a maximal effort at tumor debulking.
2. (continued from no. 1) Those patients with stage III cancer in which the largest maximal diameter of any residual tumor implant at the completion of this initial surgery is no greater than 1 cm will be defined as optimal; all others will be defined as suboptimal.
3. The histologic features of the tumor must be compatible with a primary Müllerian epithelial adenocarcinoma. Patients with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, Endometrioid adenocarcinoma, Mucinous adenocarcinoma, Undifferentiated carcinoma, Clear cell adenocarcinoma, Mixed epithelial carcinoma, Transitional cell, Malignant Brenner's Tumor, Adenocarcinoma N.O.S. Patients may have co-existing fallopian tube carcinoma in-situ so long as the primary origin of invasive tumor is ovarian, peritoneal or fallopian tube.
4. Patients must be entered no later than 12 weeks after initial surgery performed for the combined purpose of diagnosis, staging and cytoreduction.
5. Patients with measurable and non-measurable disease are eligible. Patients may or may not have cancer-related symptoms.
6. Patients in this trial may receive ovarian estrogen +/- progestin replacement therapy as indicated at the lowest effective dose(s) for control of menopausal symptoms at any time, but not progestins for management of anorexia while on protocol directed therapy.
7. Patients with an ECOG Performance Status of 0, 1, or 2.
8. Patients must have normal organ and marrow function as defined below: leukocytes >3,000/mcL; absolute neutrophil count >1,500/mcL; platelets >100,000/mcL; total bilirubin <1.5 X institutional upper limits of normal; AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal; Alkaline phosphatase (AP) <2.5 X institutional upper limit of normal; creatinine <1.5X institutional upper limit of normal OR creatinine clearance >50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent invasive epithelial ovarian, primary peritoneal or fallopian tube cancer treated with surgery only are not eligible. Patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated, new invasive epithelial ovarian, peritoneal primary or fallopian tube cancer are eligible, provided that they have not received prior chemotherapy for any ovarian tumor.
2. Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
3. Patients who have received prior chemotherapy for any abdominal or pelvic tumor including neo-adjuvant chemotherapy for their ovarian, primary peritoneal or fallopian tube cancer are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease.
4. Patients who have received any targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their epithelial ovarian or peritoneal primary cancer.
5. Patients who are currently participating or planning to participate in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study or who are receiving other investigational agents.
6. Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: Stage not greater than IB; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO Grade 3 lesions.
7. With the exception of superficial basal cell and superficial squamous (skin) cell, carcinoma in situ of the cervix and other specific malignancies as noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last five years or whose previous cancer treatment contraindicates this protocol therapy are excluded.
8. Patients with acute hepatitis or active infection that requires parenteral antibiotics.
9. Patients with serious non-healing wound, ulcer, or untreated bone fracture. This includes a history of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1. Patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations until closure.
10. Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy (in the absence of therapeutic anticoagulation), or tumor involving major vessels.
11. History of hemoptysis (>/=1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1.
12. Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study.
13. Patients with clinically significant cardiovascular disease. This includes: 1) Uncontrolled hypertension, defined as systolic > 140 mm Hg or diastolic > 90 mm Hg; 2) Myocardial infarction or unstable angina < 6 months prior to registration; 3) New York Heart Association (NYHA) Grade II or greater congestive heart failure; 4) Serious cardiac arrhythmia requiring medication. This does not include asymptomatic, atrial fibrillation with controlled ventricular rate
14. (continued from no. 13) CTCAE Grade 2 or greater peripheral vascular disease (at least brief (<24 hrs) episodes of ischemia managed non-surgically and without permanent deficit); Prior history of hypertensive crisis or hypertensive encephalopathy; Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
15. Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
16. Patients with known hypersensitivity to any component of bevacizumab
17. Patients with clinically significant proteinuria at screening as demonstrated by urine protein:creatinine (UPCR) ratio >/= 1.0 at screening. The UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection. Specifically, a UPCR of 1.0 is equivalent to 1.0 gram of protein in a 24 hour urine collection. Obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24 hour urine). Send sample to lab with request for urine protein and creatinine levels [separate requests].
18. (continued from no. 17) The lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL). The UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL).
19. Patients with or with anticipation of invasive procedures as defined below: Major surgical procedure within 28 days of initiating bevacizumab or major procedures anticipated during the course of the study. This includes, but is not limited to abdominal surgery (laparotomy or laparoscopy) prior to disease progression, such as colostomy or enterostomy reversal, interval or secondary cytoreductive surgery, or second look surgery.
20. (continued from no. 19) Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first date of bevacizumab therapy
21. Patients with ECOG Performance Grade of 3 or 4
22. Patients who are pregnant (positive pregnancy test) or nursing. Use of effective means of contraception (men and women) in subjects of child-bearing potential. To date, no fetal studies in animals or humans have been performed. The possibility of harm to a fetus is likely. Bevacizumab specifically inhibits VEGF, which is responsible for formation of new blood vessels during development, and antibodies can cross the placenta. Therefore, bevacizumab should not be administered to pregnant women.
23. (continued from no. 22) Subjects will be apprised of the large potential risk to a developing fetus. It is not known whether bevacizumab is excreted in human milk. Because many drugs are excreted in human milk, bevacizumab should not be administered to nursing women. Patients of childbearing potential must agree to use contraceptive measures during study therapy and for at least six months after completion of bevacizumab therapy.
24. Patients under the age of 18.
25. Patients who have received prior therapy with any anti-VEGF drug, including bevacizumab.
26. Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration and/or nutrition.
27. Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study.
28. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
29. Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with bevacizumab. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
30. Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-04-14 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Sood, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2010 to December 2013. All the recruitment was done in medical clinic setting.
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Carboplatin, Bevacizumab)
Started | 33
Completed | 28
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — taken off study before any treatment given | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 54 [31 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success
Description: Participants with newly diagnosed ovarian, primary peritoneal, and fallopian tube cancers treated with bevacizumab, carboplatin, and weekly paclitaxel that can tolerate at least 4 cycles of therapy regardless of delay or dose modification.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 33
Participants | 23

2. Secondary Outcome: Progression-free Survival of Optimal (RO) </= 1cm (PFS) vs Suboptimal > 1 cm
Description: Progression-Free Survival is the period from study entry until disease progression, death or date of last contact. Disease progression defined by imaging or palpation of at least a 20% increase in the sum of the LD of target lesions, the appearance of one or more new lesions, or unequivocal progression of existing nontarget lesions, the date of progression will be defined as the date such lesions were first found to be progressed by imaging or palpation. Estimated the PFS with the Kaplan-Meier product-limit estimator stratified by debulking status (optimal, sub-optimal).The Cox proportional hazards regression model to assess the association of gene expression and cytokines with PFS.
Time Frame: 2 years
Population: 3 participants were not evaluable due to post surgical complications.
Measure: Median (Full Range); unit: Number of months
Arm/Group | Treatment (Paclitaxel, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 30
Number of months
  Optimal (no residual): number analyzed (Participants) | 16
  Optimal (no residual) | 22.4 [5.4 to 32.8]
  Optimal (<1 cm): number analyzed (Participants) | 9
  Optimal (<1 cm) | 16.9 [4.8 to 30.5]
  Suboptimal (>1 cm): number analyzed (Participants) | 5
  Suboptimal (>1 cm) | 16.9 [3.9 to 19.2]
Statistical Analysis 1: Comparison: Treatment (Paclitaxel, Carboplatin, Bevacizumab); Participants for optimal ≤ 1 cm; Test type: Superiority; p = 0.33, t-test, 2 sided; Hazard Ratio (HR) = 1.71, 95% CI 2-sided [0.58 to 4.98]
Statistical Analysis 2: Comparison: Treatment (Paclitaxel, Carboplatin, Bevacizumab); suboptimal > 1 cm; Test type: Superiority; p = 0.04, t-test, 2 sided; Hazard Ratio (HR) = 3.75, 95% CI 2-sided [1.05 to 13.34]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the start of the study until 30 days after the last dose of study medication taken, up to a maximum of 32.8 months
Arm/Group | Treatment (Paclitaxel, Carboplatin, Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 3/33
Other Adverse Events (participants affected / at risk) | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Bevacizumab) (N=33)
Wound dehisence (Injury, poisoning and procedural complications) | 1
Neutropenia (Investigations) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Bevacizumab) (N=33)
Anemia (Blood and lymphatic system disorders) | 16
Neutropenia (Investigations) | 16
Decrease Platelets (Investigations) | 9
Leukopenia (Investigations) | 11
Fatigue (General disorders) | 23
Constipation (Gastrointestinal disorders) | 20
Diarrhea (Gastrointestinal disorders) | 8
Pain (General disorders) | 18
Alopecia (Skin and subcutaneous tissue disorders) | 23
Mucositis (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 14
Neuropathy (Nervous system disorders) | 11
Liver Enzymes (Investigations) | 4
Rash (Skin and subcutaneous tissue disorders) | 8
Nail disorder (Infections and infestations) | 3
Infection (Infections and infestations) | 3
Flushing (Vascular disorders) | 2
Insomnia (Psychiatric disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Anxiety (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT01097746/Prot_SAP_000.pdf